CLINICAL TRIAL: NCT05992116
Title: The Prevalence of Iron Deficiency in Patients With Heart Failure (HFrEF and HFmrEF) in a Middle Eastern Population
Brief Title: Iron Deficiency in Patients With Heart Failure and Reduced and Mildly Reduced Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: RT.IrnDefHFr.mr.EF.Jo001
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-03

CONDITIONS: Iron Deficiency; Heart Failure With Reduced Ejection Fraction; Heart Failure With Mildly Reduced Ejection Fraction
Keywords: Iron deficiency; Heart failure; Heart failure with reduced ejection fraction; Heart failure with mildly reduced ejection fraction
MeSH Terms: conditions — Iron Deficiencies; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A significant percentage of patients with heart failure and reduced ejection fraction (HFrEF) or mildly reduced ejection fraction (HFmrEF) have iron deficiency who are symptomatic. This is independently associated with bad quality of life, low functional capacity, lower quality of, life and increased mortality. The prevalence of iron deficiency in HFrEF and HFmrEF patients in Jordan has not been studied in the past.

DETAILED DESCRIPTION:
The prevalence of chronic heart failure among the industrialized countries is 1-3%, and can exceed 30% in the elderly population. As the population ages, there is an increase in the number of co-morbidities among heart failure patients. These comorbidities are associated with an increase in major adverse cardiac events (MACE), cost, and complexity of care. Iron deficiency is one of the most common comorbidities occurring in patients with heart failure. Its prevalence can be as high as 59%, even if patients are non-anemic[4]. Iron deficiency in heart failure can lead to an impaired exercise capacity, a decreased quality of life and an increased risk of hospitalizations and mortality regardless of anemia. The relationship between the severity of iron deficiency and the prognosis is a linear one, with increased severity being associated with increased mortality.

Intravenous iron treatment has been shown to improve the quality of life, with an increased exercise capacity and a reduced risk for hospitalizations. The prevalence of iron deficiency in HFrEF and HFmrEF patients in Middle Eastern population has not been studied. We suspect a higher prevalence compared to Western populations especially in women.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with ejection fraction <59% (including those with with reduced ejection fraction of ≤40%, or mildly reduced EF (41-49%)) within the last 2 years.
* NYHA class II-IV.
* Able and willing to provide oral informed consent.

Exclusion Criteria:

* Age<18 years.
* Acute coronary syndrome.
* Known cases of iron overload (e.g. hemochromatosis); known cases of anemia due to other causes.
* Oral or intravenous iron supplements within the previous 3 months; erythropoietin stimulating agents or blood transfusion within the last 6 months.
* Active clinically relevant bleeding in the investigator's opinion.
* Patients with chronic inflammatory conditions (e.g. rheumatoid arthritis; Crohn's disease, etc.); active infection; and decompensated liver disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers who are adults (18 years of age or older) who have heart failure and an ejection fraction <50%.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Iron deficiency | From date of study enrollment until the date of first documented diagnosis of iron deficiency up to 2 weeks.
  A serum ferritin level of <100 ng/ml, or a serum ferritin level of 100-299 ng/ml with a TSAT of < 20% confirms the diagnosis of iron deficiency, regardless of the HB level. TSAT is calculated by the following formula: Serum iron/ TIBC *100.

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Tabbalat, Study Chair — Abdali Hospital
Locations (1):
- Abdali Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Emails and via WhatsApp group to local cardiologists to introc=duce the study to them
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After clinicaltrials.gov sends us an identifier number